CLINICAL TRIAL: NCT03233373
Title: Thermal Imaging as a Potential Diagnostic Tool of Nasal Airflow. A Pilot Study.
Brief Title: Thermal Imaging as a Potential Diagnostic Tool of Nasal Airflow
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Howard Stupak, Director, Department of Otolaryngology at Jacobi Medical Center / Associate Professor Department of Otorhinolaryngology - Albert Einstein College of Medicine, New York City Health and Hospitals Corporation
Other Study IDs: 2017-8248
Record Dates: First submitted 2017-07-17; First posted 2017-07-28 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Nasal Airway Obstruction
Keywords: Nasal Airway Obstruction; Devices; Imaging, Diagnostic; Computer-Assisted Image Processing; Thermal Analysis, Differential
MeSH Terms: conditions — Nasal Obstruction; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Otolaryngology Clinic Patients: Healthy subjects with no present complaints of nasal obstructions. Patients visiting the clinic, once consented, will be asked which nostril they breathe better from. They will then be asked to perform 3-4 normal respiration cycles through their nose which will be recorded using our thermal imaging device, the Seek CompactPro thermal imager
  Interventions: Device: Seek CompactPro thermal imager

INTERVENTIONS:
Device: Seek CompactPro thermal imager — A device with image/video recording capability, it is non-invasive and only relies on infrared emissions from heat sources (the patient).

SUMMARY:
Currently, there are no tools that can measure nasal airflow in an objective manner that is non-invasive to the patient. This clinical study aims to address this by evaluating the use of thermal imaging as a diagnostic tool for measuring nasal airflow.

Proper airflow cools the nasal airway as it passes--obstructions or narrowed airways hinder flow and results in elevated temperatures along the airway and nasal tissue. It is this elevation in temperature, or more specifically, loss of cooling, that we hypothesize to be measurable with thermal imaging. Participants in this study will be asked to perform 3-4 nasal breathing cycles which will be recorded by the thermal imager.

DETAILED DESCRIPTION:
Currently there's no non-invasive, objective method for measuring nasal airflow. The current standard, the NOSE score is an inaccurate measure of physiology (it is subjective). There is a considerable amount of data that demonstrates that the nasopharyngeal airway is the preferred ventilatory pathway for breathing at rest and during sleep. Finding a reliable measurement modality is important in light of this. The primary goal of this study is to evaluate a novel approach to measuring nasal airflow in thermal imaging. Previous studies show that higher temperatures of the nasal mucosa are related to decreased patency. The investigators hypothesize that reduced or obstructed airflow leads to the loss of the cooling oscillatory cycle present in normal nasal respiration. The investigators believe this diminished or absent cycle may be detectable via thermal imaging due to predicted elevation of mucosal temperatures (or loss of the cooling gradient). Other methods in the past aimed at measuring temperature changes introduced error due to their invasiveness (irritation of the mucosa lead to higher baseline oscillatory cycles). This is no longer an issue as the thermal imager requires no physical contact with the patient to function.

There are several methods for measuring nasal patency that have been described throughout the literature. These include objective measurements such as acoustic rhinometry and rhinomanometry, as well as subjective measurements such as the Sino-Nasal Outcome Test and Nasal Obstruction Symptom Evaluation (NOSE) questionnaires. More recently, snap-on thermal imaging devices that take advantage of the processing power and high resolution of modern phones have surfaced leading to lower costs for highly-sensitive devices that we aim to use for measuring nasal airflow. The non-invasive nature of using thermal devices may lead to more accurate, objective measurements of nasal airflow as a previous study demonstrated that tactile irritation from other devices increase the mucosal temperature impeding measurement. (Bailey et al.). Other studies documented that improved sensation of nasal airflow is associated with cooler mucosal temperatures and that increased patency of the nasal passage is related to lower temperatures as well (and the opposite, decreased patency to increased temperatures). (Willatt et al.) We hypothesize that nasal airflow obstruction (NAO) leads to the loss of the cooling oscillatory cycle present in normal nasal respiration which we can detect via thermal imaging due to predicted elevation of mucosal temperatures.

ELIGIBILITY:
Inclusion Criteria:

- All adult patients presenting to the Jacobi Medical Center otolaryngology clinic

Exclusion Criteria:

* Patients under the age of 18
* Patients who recently used any nasal decongestants the day of measurement
* Patients with an active infection such as sinusitis
* Patients with anatomical abnormalities such a severe septal deviation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy patients with no present congestion or complaints of nasal obstruction.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Minimum temperature in centigrade of patient's reported better (more patent) and worse (less patent) nasal airway | through study completion, an average of 1 year
  From recorded thermal imaging of nasal respiration cycles of both nostrils (nasal airways)

SECONDARY OUTCOMES:
Area of cooling of patient's reported better (more patent) and worse (less patent) nasal airway | through study completion, an average of 1 year
  From recorded thermal imaging of nasal respiration cycles of both nostrils (nasal airways)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Stupak, MD, Principal Investigator — NYCHHC, Albert Einstein College of Medicine
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey RS, Casey KP, Pawar SS, Garcia GJ. Correlation of Nasal Mucosal Temperature With Subjective Nasal Patency in Healthy Individuals. JAMA Facial Plast Surg. 2017 Jan 1;19(1):46-52. doi: 10.1001/jamafacial.2016.1445. PMID 27918749
- [Background] Roblin DG, Eccles R. Normal range for nasal partitioning of airflow determined by nasal spirometry in 100 healthy subjects. Am J Rhinol. 2003 Jul-Aug;17(4):179-83. PMID 12962185
- [Background] Tsounis M, Swart KM, Georgalas C, Markou K, Menger DJ. The clinical value of peak nasal inspiratory flow, peak oral inspiratory flow, and the nasal patency index. Laryngoscope. 2014 Dec;124(12):2665-9. doi: 10.1002/lary.24810. Epub 2014 Jul 30. PMID 25073629
- [Background] Willatt DJ. Continuous infrared thermometry of the nasal mucosa. Rhinology. 1993 Jun;31(2):63-7. PMID 8362171
- [Background] Willatt DJ, Jones AS. The role of the temperature of the nasal lining in the sensation of nasal patency. Clin Otolaryngol Allied Sci. 1996 Dec;21(6):519-23. doi: 10.1111/j.1365-2273.1996.tb01102.x. PMID 9118573
- [Background] Zhao K, Blacker K, Luo Y, Bryant B, Jiang J. Perceiving nasal patency through mucosal cooling rather than air temperature or nasal resistance. PLoS One. 2011;6(10):e24618. doi: 10.1371/journal.pone.0024618. Epub 2011 Oct 13. PMID 22022361
- [Background] Chaaban M, Corey JP. Assessing nasal air flow: options and utility. Proc Am Thorac Soc. 2011 Mar;8(1):70-8. doi: 10.1513/pats.201005-034RN. PMID 21364224